CLINICAL TRIAL: NCT04662372
Title: Functional Neurological Disorders in Patients Admitted in Stroke Units: Clinical Profile et and 6 Months Follow-up
Brief Title: Functional Neurological Disorders in Patients Admitted in Stroke Units
Acronym: NEUROFON
Status: Active, not recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SBY_2020_1
Record Dates: First submitted 2020-10-09; First posted 2020-12-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Functional Neurological Disorders
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients
  Interventions: Other: Description

INTERVENTIONS:
Other: Description — description of the cognitive and behavioral profile of stroke mimics patients, without evidence of neurological disease.

SUMMARY:
Functional neurological disorders are an important subgroup of patients with stroke mimics admitted to stroke unit.Their clinical profile and outcome are poorly known. The goal of this study is to describe the cognitive and behavioral profile of stroke mimics patients, without evidence of neurological disease.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Patients admitted in stroke unit for a neurological deficit, without evidence of neurovascular or othe neurological disease.
* NIHSS ≥ 1 at time of admission
* Informed and consent patient to study
* Health insured

Exclusion Criteria:

* Patient receiving legal protection
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in stroke unit for a neurological deficit, without evidence of neurovascular or othe neurological disease
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Patient characteristics | 3 months
  Cognitive/behavioural characteristics of patients assessed for stroke using the National Institute of Health Stroke Score ranging from 0 to 42 (0: no stroke; 1-4: minor stroke; 5-15: moderate stroke; moderate to severe stroke; 21-42: severe stroke)

SECONDARY OUTCOMES:
symptoms of patients | 3 and 6 months
  Description of symptoms at 3 and 6 months after transition in stroke unit

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Fondation Adolphe de Rothschild, Paris, Paris, France